CLINICAL TRIAL: NCT06389695
Title: Pharmacokinetics, Biodistribution, Radiation Dose and Safety Study of a Single Dose of Gallium [68Ga]-NYM032 Injection Prepared by Kit for the Preparation of the 68Ga-NYM032 Injection in Patients With Prostate Cancer
Brief Title: Pharmacokinetics, Biodistribution, Radiation Dose and Safety Study of 68Ga-NYM032 in Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Norroy Bioscience Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP-2023-03; NYM032D01 (Other: National Medical Products Administration)
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-NYM032 injection (Experimental)
  Interventions: Drug: 68Ga-NYM032 injection

INTERVENTIONS:
Drug: 68Ga-NYM032 injection — The radiation dose is about 3-6 mCi for a single patient.Using a syringe to withdraw 68Ga-NYM032 injection, the dose will be administered via an intravenous injection and the injection time will be about 45-60 seconds.

SUMMARY:
68Ga-NYM032 is a PSMA-targeting small-molecular radiotracer for PET/CT imaging of prostate cancer, which is needed for clinical trial to be conducted

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed prostate cancer;
2. Age range from 18 to 75 years old (including 18 and 75 years old);
3. ECOG score of 0 or 1;
4. Expected life ≥ 6 months；
5. The subjects agree to take effective contraceptive measures during the study period and for at least three months after the diug administration;
6. The subjects are able to maintain good communication with the researchers；understand and follow the requirements of this study and sign an informed consent form before the start of relevant research operations.

Exclusion Criteria:

1. Known or suspected to be allergic to the investigational drug or any of its components;
2. Accepting other investigational drugs upon enrollment, or within 5 biological half-lives of the drug at enrollment, or within 30 days after its last administration, whichever is longer;
3. Those who have used any radioactive therapy medication within 90 days before investigational drug administration, or have received any radioactive diagnostic medication within 3 days before investigational drug administration;
4. Planned androgen deprivation therapies use, any therapeutic intervention for the prostate cancer and use of folate supplements during the study;
5. Plan to arrange surgery and other invasive interventions within 2 days after the injection of the investigational drug；
6. Ongoing toxicity >grade l from previous standard or investigational therapies；
7. Patients with active infections during screening;
8. Those who have no guarantee of being able to lie down quietly in the examination cabin during a PET examination, or those who suffer from claustrophobia and cannot cooperate in a PET examination:
9. Other situations where the researchers believe that the subject is not suitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 5 days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Peking Union Medical College Hospital, Beijing

REFERENCES:
- [Derived] Fu H, He H, Wang Y, Li W, Luo Y, Chen L, Mi Y, Sun C, Mao Y, Yu C. Preliminary evaluation of a novel PSMA-targeting radiopharmaceutical [68Ga]Ga/[177Lu]Lu-NYM032 for theranostic use in prostate cancer. Eur J Nucl Med Mol Imaging. 2025 Apr;52(5):1671-1684. doi: 10.1007/s00259-024-07046-5. Epub 2025 Jan 2. PMID 39745526